CLINICAL TRIAL: NCT00003381
Title: Quality of Life and Cost Analysis of a Prospective Randomized Phase III Trial Comparing Trimodality Therapy to Surgery Alone for Esophageal Cancer [Companion to CALGB-9781]
Brief Title: Quality of Life Assessment of Patients Receiving Treatment for Esophageal Cancer [Companion to CALGB-9781]
Status: Terminated | Type: Observational
Why Stopped: companion study to CALGB-9781 which closed administratively due to poor accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-9870; CDR0000066376 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Questionnaires that measure quality of life during treatment may improve the ability to plan treatment for patients with esophageal cancer.

PURPOSE: This clinical trial is studying the quality of life in patients receiving treatment for esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the quality of life of patients with esophageal cancer randomized on protocol CALGB C9781 to treatment with surgery alone vs trimodal therapy combining preoperative chemotherapy and radiation therapy in addition to surgery. II. Examine the incremental cost and cost effectiveness of preoperative chemotherapy and radiation therapy in the treatment of esophageal cancer. III. Examine the incremental cost per quality-adjusted life year (QALY) of preoperative chemotherapy and radiation therapy in the treatment of esophageal cancer.

OUTLINE: This is a companion study to CALGB C9781, a phase III randomized study. Prior to treatment on CALGB C9781, patients complete forms assessing quality of life, psychological functioning, specific areas of dysfunction, resource use, and time lost from work; subsequent assessments are completed by telephone interview at 1, 2, 6, 12, 18, and 24 months after the initiation of study treatment, regardless of disease status (patients with hearing impairment and those speaking only a translatable foreign language may mail responses). Patients also keep a diary of medical resource utilization at sites other than the treating institution.

ELIGIBILITY:
1. Patients with histologically documented untreated squamous cell carcinoma or adenocarcinoma of the thoracic esophagus (below 20 cm) or gastroesophageal junction and with less than 2cmdistal spread into the gastric cardia eligible for C9781.
2. There could be no evidence of distant metastatic disease by history and physical examination; upper endoscopy with biopsy, computed tomography (CT) of the chest and upper abdomen, and pulmonary function studies were all required.
3. Tumors had to be considered surgically resectable (T1-3, NX), including regional thoracic lymph node (N1) metastases.
4. Patients with supraclavicular lymph nodes measuring ≤1.5 cm by CT (not palpable) were eligible, as were patients with lymph node metastases to levels 15 to 20 (predominantly celiac axis and paracardial nodes) ≤ 1.5 cm by CT.
5. Patients could not have previously received chemotherapy or radiation therapy for this tumor or any radiation therapy that would overlap the radiation fields required for this malignancy. Patients with previous malignancies were eligible if more than 5 years had elapsed from diagnosis without evidence of tumor recurrence.
6. There could be no other serious illness that would limit survival to less than 2 years, or psychiatric condition that would prevent compliance with treatment or informed consent.
7. Patients with uncontrolled or severe cardiovascular disease, pulmonary disease, or active infections were excluded, as were pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer eligible to participate in C9781.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 1998-07; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the quality of life of patients | Up to 3 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: David G. Pfister, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (44):
- United States (44):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia